CLINICAL TRIAL: NCT04819295
Title: Barriers, Facilitators, and Preferences Regarding Depression Treatment From the Perspectives of Latinx Adolescents, Parents, and Healthcare Providers
Brief Title: Latinx Teen Depression Treatment Study
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00107485
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-03

CONDITIONS: Depression
Keywords: Latinx adolescents; psychotherapy; Focus groups
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Latinx Adolescents
- Parents of Latinx Adolescents
- Healthproviders

SUMMARY:
The purpose of this study is determine facilitators of and barriers to receiving evidence-based psychotherapy for depression for Latinx adolescents from multiple stakeholder perspectives.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13-17
* self-identify as Hispanic/Latinx
* diagnosed with Major Depressive Disorder or Persistent Depressive Disorder/Dysthymia
* referred to psychotherapy or prescribed medication for depression.

Healthcare providers:

* Self-identify as regularly providing clinical care to Latinx adolescents with depression
* be in a role in which they can refer to or provide depression treatment.

Exclusion Criteria:

* Teens will be excluded if they are experiencing intense psychological distress or imminent thoughts of suicide or have any condition in which, in the opinion of the investigator, precludes the study team from obtaining informed assent of the teen

Ages: 13 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Latnix adolescents and their parents, including healthcare providers who are involved in psychotherapy treatments.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of preferences for depression treatment generated from focus groups | Baseline

SECONDARY OUTCOMES:
Number of barriers to depression treatment among Latinx Adolescents from focus groups | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Allison Stafford, Ph.D, Principal Investigator — Duke University
Locations (1):
- DUSON, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No